CLINICAL TRIAL: NCT00959946
Title: A Phase 1/2, Open-Label Study Of Bosutinib Administered In Combination With Capecitabine In Subjects With Solid Tumor And ErbB2 Negative Locally Advanced Or Metastatic Breast Cancer
Brief Title: Study Of Bosutinib With Capecitabine In Solid Tumors And Locally Advanced Or Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3160A6-2208; B1871011
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Results first posted 2013-02-22 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-01

CONDITIONS: Advanced Breast Cancer (Parts 1 and 2); Advanced Pancreatic Cancer (Part 1); Advanced Colorectal Cancer (Part 1); Advanced Cholangiocarcinoma (Part 1); Advanced Glioblastoma Multiforme (Part 1)
Keywords: Phase 1/2; 2-part study; bosutinib and capecitabine
MeSH Terms: interventions — bosutinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): In part 1 (phase 1), ascending and descending multiple oral doses of bosutinib + capecitabine. Doses in part 1 include capecitabine 750 mg/m2 BID on days 1-14 + bosutinib 200 mg QD; capecitabine 625 mg/m2 BID on days 1-14 + bosutinib 300 mg QD. Depending on safety, capecitabine can also be administered at 1000 mg/m2 BID and bosutinib can be administered at 200 mg/m2 QD. The MTD of the combination treatment determined from part 1, will be administered in part 2 (phase 2).
  Interventions: Drug: Bosutinib; Drug: Capecitabine

INTERVENTIONS:
Drug: Bosutinib — Doses in part 1 include bosutinib 200 mg QD; bosutinib 300 mg QD. Depending on safety bosutinib can be administered at 200 mg/m2 QD. The MTD of the combination treatment determined from part 1, will be administered in part 2 (phase 2).
Drug: Capecitabine — Doses in part 1 include capecitabine 750 mg/m2 BID on days 1-14; capecitabine 625 mg/m2 BID on days 1-14. Depending on safety, capecitabine can also be administered at 1000 mg/m2 BID. The MTD of the combination treatment determined from part 1, will be administered in part 2 (phase 2).

SUMMARY:
This is a research study in 2 parts assessing the following parameters of the combination of the study drug called bosutinib, and a drug called capecitabine: the safety, how well the subject's body handles the study drug, and preliminary anti-tumor activity as treatment for different types of cancers in part 1, and breast cancer only in part 2.

In part 1, subjects will receive bosutinib and capecitabine daily at different dose levels of each drug in order to determine the highest tolerated dose of the combination study treatment. In part 2, subjects will receive bosutinib and capecitabine at this highest tolerated dose to see how well the study treatment works to treat breast cancer. In addition, genetic research testing (research analyses involving genes and gene products) will be performed on biological samples from subjects.

DETAILED DESCRIPTION:
The study was prematurely discontinued following Part 1 evaluation, when the sponsor concluded that further translational biomarker analyses were needed to better define the breast tumor biomarkers that predict sensitivity to Src family kinase inhibitors. Thus the Sponsor made a determination to stop the study after Part 1 as communicated to investigators on 02Dec2010 . No subjects were enrolled into Part 2 of this study. The study was not terminated due to safety reasons.

ELIGIBILITY:
Inclusion Criteria:

Part 1:

* Ages eligible for study: 18 years or older.
* Male and female.
* Confirmed pathologic diagnosis of advanced breast cancer or pancreatic cancer or colorectal cancer or cholangiocarcinoma or glioblastoma not curable with available therapies, for whom bosutinib plus capecitabine is a reasonable treatment option.

Part 2:

* Ages eligible for study: 18 years or older.
* Female.
* Confirmed pathologic diagnosis of locally advanced or metastatic breast cancer, or loco-regional recurrent breast cancer that is not amenable to curative treatment with surgery or radiotherapy.
* Documented ER+ and/or PgR+/erbB2- or ER-/PgR-/erbB2- tumor based upon recently analyzed biopsy.

Exclusion Criteria:

Part 1:

* Prior bosutinib, or any other prior Src inhibitor.
* Prior chemotherapy with capecitabine or 5-FU for the treatment of metastatic disease is allowed unless patient stopped therapy for toxicity.

Part 2:

* Prior bosutinib, or any other prior Src inhibitor prior chemotherapy with capecitabine or 5-FU for the treatment of metastatic disease.
* Prior chemotherapy with capecitabine or 5-FU for adjuvant chemotherapy within the past 12 months.
* erbB2+ breast cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- United States (2):
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Detroit, Michigan
- Pfizer Investigational Site, Adelaide, South Australia, Australia
- Pfizer Investigational Site, Edegem, Belgium
- Pfizer Investigational Site, Saint-Herblain, France
- Pfizer Investigational Site, Hong Kong, Hong Kong
- Pfizer Investigational Site, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Isakoff SJ, Wang D, Campone M, Calles A, Leip E, Turnbull K, Bardy-Bouxin N, Duvillie L, Calvo E. Bosutinib plus capecitabine for selected advanced solid tumours: results of a phase 1 dose-escalation study. Br J Cancer. 2014 Nov 25;111(11):2058-66. doi: 10.1038/bjc.2014.508. Epub 2014 Oct 7. PMID 25290090
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3160A6-2208&StudyName=Study%20Of%20Bosutinib%20With%20Capecitabine%20In%20Solid%20Tumors%20And%20Locally%20Advanced%20Or%20Metastatic%20Breast%20Cancer

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was pre-maturely terminated after part 1 (safety lead-in phase) of study and hence, planned treatments of part 2, Bosutinib 300 milligram (mg) + Capecitabine 1000 mg/square meter (mg/m^2) (Part 2): estrogen receptor positive (ER+) and Bosutinib 300 mg+Capecitabine 1000 mg/m^2 (Part 2): estrogen receptor negative (ER-), were not administered.
Groups:
- Bosutinib 200 mg + Capecitabine 625 mg/m^2 (Part 1): Bosutinib 200 mg tablet orally once daily in a 21-day cycle along with capecitabine 625 mg/m^2 tablet orally twice daily from Day 1 to 14, followed by 7 days off treatment in a 21-day cycle. Treatment was continued until disease progression, unacceptable toxicity, or withdrawal of consent.
- Bosutinib 200 mg + Capecitabine 750 mg/m^2 (Part 1): Bosutinib 200 mg tablet orally once daily in a 21-day cycle along with capecitabine 750 mg/m^2 tablet orally twice daily from Day 1 to 14, followed by 7 days off treatment in a 21-day cycle. Treatment was continued until disease progression, intolerable toxicity, or withdrawal of consent.
- Bosutinib 200 mg + Capecitabine 1000 mg/m^2 (Part 1): Bosutinib 200 mg tablet orally once daily in a 21-day cycle along with capecitabine 1000 mg/m^2 tablet orally twice daily from Day 1 to 14, followed by 7 days off treatment in a 21-day cycle. Treatment was continued until disease progression, intolerable toxicity, or withdrawal of consent.
- Bosutinib 300 mg + Capecitabine 625 mg/m^2 (Part 1): Bosutinib 300 mg tablet orally once daily in a 21-day cycle along with capecitabine 625 mg/m^2 tablet orally twice daily from Day 1 to 14, followed by 7 days off treatment in a 21-day cycle. Treatment was continued until disease progression, intolerable toxicity, or withdrawal of consent.
- Bosutinib 300 mg + Capecitabine 750 mg/m^2 (Part 1): Bosutinib 300 mg tablet orally once daily in a 21-day cycle along with capecitabine 750 mg/m^2 tablet orally twice daily from Day 1 to 14, followed by 7 days off treatment in a 21-day cycle. Treatment was continued until disease progression, intolerable toxicity, or withdrawal of consent.
- Bosutinib 300 mg + Capecitabine 1000 mg/m^2 (Part 1): Bosutinib 300 mg tablet orally once daily in a 21-day cycle along with capecitabine 1000 mg/m^2 tablet orally twice daily from Day 1 to 14, followed by 7 days off treatment in a 21-day cycle. Treatment was continued until disease progression, intolerable toxicity, or withdrawal of consent.
- Bosutinib 400 mg + Capecitabine 750 mg/m^2 (Part 1): Bosutinib 400 mg tablet orally once daily in a 21-day cycle along with capecitabine 750 mg/m^2 tablet orally twice daily from Day 1 to 14, followed by 7 days off treatment in a 21-day cycle. Treatment was continued until disease progression, intolerable toxicity, or withdrawal of consent.
- Bosutinib 400 mg + Capecitabine 1000 mg/m^2 (Part 1): Bosutinib 400 mg tablet orally once daily in a 21-day cycle along with capecitabine 1000 mg/m^2 tablet orally twice daily from Day 1 to 14, followed by 7 days off treatment in a 21-day cycle. Treatment was continued until disease progression, intolerable toxicity, or withdrawal of consent.
Period: Overall Study
Arm/Group | Bosutinib 200 mg + Capecitabine 625 mg/m^2 (Part 1) | Bosutinib 200 mg + Capecitabine 750 mg/m^2 (Part 1) | Bosutinib 200 mg + Capecitabine 1000 mg/m^2 (Part 1) | Bosutinib 300 mg + Capecitabine 625 mg/m^2 (Part 1) | Bosutinib 300 mg + Capecitabine 750 mg/m^2 (Part 1) | Bosutinib 300 mg + Capecitabine 1000 mg/m^2 (Part 1) | Bosutinib 400 mg + Capecitabine 750 mg/m^2 (Part 1) | Bosutinib 400 mg + Capecitabine 1000 mg/m^2 (Part 1)
Started | 2 | 4 | 4 | 5 | 4 | 9 | 2 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 4 | 4 | 5 | 4 | 9 | 2 | 2
Not completed — Adverse Event | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Disease Progression | 2 | 4 | 2 | 4 | 4 | 6 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bosutinib 200 mg + Capecitabine 625 mg/m^2 (Part 1) | Bosutinib 200 mg + Capecitabine 750 mg/m^2 (Part 1) | Bosutinib 200 mg + Capecitabine 1000 mg/m^2 (Part 1) | Bosutinib 300 mg + Capecitabine 625 mg/m^2 (Part 1) | Bosutinib 300 mg + Capecitabine 750 mg/m^2 (Part 1) | Bosutinib 300 mg + Capecitabine 1000 mg/m^2 (Part 1) | Bosutinib 400 mg + Capecitabine 750 mg/m^2 (Part 1) | Bosutinib 400 mg + Capecitabine 1000 mg/m^2 (Part 1) | Total
Number analyzed (Participants) | 2 | 4 | 4 | 5 | 4 | 9 | 2 | 2 | 32
Age Continuous [Mean (Standard Deviation); unit: Years] | 53.0 (4.24) | 56.8 (16.32) | 67.3 (10.05) | 63.0 (8.43) | 56.0 (8.45) | 63.8 (5.49) | 51.5 (6.36) | 61.5 (4.95) | 60.7 (9.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 4 | 3 | 4 | 1 | 1 | 18
  Male | 0 | 3 | 2 | 1 | 1 | 5 | 1 | 1 | 14

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) - Part 1
Description: The MTD contour is defined as the dose combinations that achieve a toxicity rate (dose-limiting toxicity [DLT] rate) of less than (<) 1/3. The observed toxicity rates for all the reporting groups (to which at least 1 cohort of participants was allocated) was estimated by calculating the proportion of DLTs observed in the first 21 days of treatment at those reporting groups. DLT includes grade (Gr) 3/4 nausea, vomiting, diarrhea, or asthenia more than 3 days, Gr 4 hematologic toxicities, delayed study treatment administration due to dose toxicities by more than 3 weeks. Pre-defined criterion for MTD: if a higher dose level of capecitabine existed such that the same dose level of bosutinib had a DLT rate of <1/3, no MTD was recommended for that capecitabine dose and if even the lowest dose of bosutinib achieved a toxicity rate of greater than (>) 1/3, no MTD was recommended for that capecitabine dose level.
Time Frame: Part 1 Baseline up to Day 21
Population: DLT evaluable population included all participants who received at least 14 doses of bosutinib and at least 10 doses of capecitabine in the first 21 days of treatment or had experienced a DLT within the first 21 days of treatment. N (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Number; unit: mg
Groups:
- Bosutinib + Capecitabine 625 mg/m^2: Bosutinib 200 mg, or 300 mg, tablet administered orally once daily in a 21-day cycle. Capecitabine 625 mg/m^2 tablet administered orally twice daily from Day 1 to 14, followed by 7 days off treatment in a 21-day cycle. Treatment was continued until disease progression, intolerable toxicity, or withdrawal of consent.
- Bosutinib + Capecitabine 750 mg/m^2: Bosutinib 200 mg, 300 mg, or 400 mg tablet administered orally once daily in a 21-day cycle. Capecitabine 750 mg/m^2 tablet administered orally twice daily from Day 1 to 14, followed by 7 days off treatment in a 21-day cycle. Treatment was continued until disease progression, intolerable toxicity, or withdrawal of consent.
- Bosutinib + Capecitabine 1000 mg/m^2: Bosutinib 200 mg, 300 mg, or 400 mg tablet administered orally once daily in a 21-day cycle. Capecitabine 1000 mg/m^2 tablet administered orally twice daily from Day 1 to 14, followed by 7 days off treatment in a 21-day cycle. Treatment was continued until disease progression, intolerable toxicity, or withdrawal of consent.
Arm/Group | Bosutinib + Capecitabine 625 mg/m^2 | Bosutinib + Capecitabine 750 mg/m^2 | Bosutinib + Capecitabine 1000 mg/m^2
Number analyzed (Participants) | 6 | 10 | 8
mg | NA — MTD was not achieved since none of the participants experienced dose-limiting toxicity. | NA — Bosutinib 400 mg + Capecitabine 750 mg/m^2 had DLT >1/3, and both Bosutinib 300 mg + Capecitabine 1000 mg/m^2 and Bosutinib 300 mg + Capecitabine 750 mg/m^2 had DLT <1/3, hence no MTD for Capecitabine 750 mg/m^2 as per pre-defined criterion. | 300

2. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs) - Part 1
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Part 1 Baseline up to 28 days after last dose of study treatment
Population: Safety population: included participants who received at least 1 dose of the study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Bosutinib 200 mg + Capecitabine 625 mg/m^2 (Part 1) | Bosutinib 200 mg + Capecitabine 750 mg/m^2 (Part 1) | Bosutinib 200 mg + Capecitabine 1000 mg/m^2 (Part 1) | Bosutinib 300 mg + Capecitabine 625 mg/m^2 (Part 1) | Bosutinib 300 mg + Capecitabine 750 mg/m^2 (Part 1) | Bosutinib 300 mg + Capecitabine 1000 mg/m^2 (Part 1) | Bosutinib 400 mg + Capecitabine 750 mg/m^2 (Part 1) | Bosutinib 400 mg + Capecitabine 1000 mg/m^2 (Part 1)
Number analyzed (Participants) | 2 | 4 | 4 | 5 | 4 | 9 | 2 | 2
Percentage of Participants
  AEs | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0
  SAEs | 0.0 | 50.0 | 50.0 | 40.0 | 0.0 | 33.3 | 0.0 | 50.0

3. Primary Outcome: Percentage of Participants With Objective Response - Part 2
Description: Percentage of participants with objective response based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST v1.0). Confirmed responses are those that persist on repeat imaging study at least 4 weeks after initial documentation of response. CR is defined as the disappearance of all lesions (target and/or non target). PR are those with at least 30 percent (%) decrease in the sum of the longest dimensions (LDs) of the target lesions taking as a reference the baseline sum LDs.
Time Frame: Part 2 Baseline, every 6 weeks up to 2 to 6 weeks after last dose
Population: Data was not analyzed because the study was prematurely terminated due to unfavorable risk benefit ratio of the study treatment.
Groups:
- Bosutinib 300 mg + Capecitabine 1000 mg/m^2 (Part 2): ER+: Bosutinib 300 mg orally once daily in a 21-day cycle along with capecitabine 1000 mg/m^2 orally twice daily from Day 1 to 14, followed by 7 days off treatment in a 21-day cycle, until disease progression, intolerable toxicity, or withdrawal of consent in participants with locally advanced or metastatic breast cancer having estrogen receptor positive (ER+) and/or progesterone receptor positive (PgR+) and human epidermal growth factor receptor 2 negative (erbB2-).
- Bosutinib 300 mg + Capecitabine 1000 mg/m^2 (Part 2): ER-: Bosutinib 300 mg orally once daily in a 21-day cycle along with capecitabine 1000 mg/m^2 orally twice daily from Day 1 to 14, followed by 7 days off treatment in a 21-day cycle, until disease progression, intolerable toxicity, or withdrawal of consent in participants with locally advanced or metastatic breast cancer having estrogen receptor negative (ER-) and/or progesterone receptor negative (PgR-) and human epidermal growth factor receptor 2 negative (erbB2-).
Arm/Group | Bosutinib 300 mg + Capecitabine 1000 mg/m^2 (Part 2): ER+ | Bosutinib 300 mg + Capecitabine 1000 mg/m^2 (Part 2): ER-
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Best Overall Response - Part 1
Description: Best overall response based on investigator's disease status assessment. CR: disappearance of all lesions. PR: at least 30% decrease in sum of LDs of target lesions taking as reference baseline sum LDs. Progressive disease (PD): at least 20% increase in sum of LD of target lesions taking as a reference smallest sum of the recorded LDs since treatment start, or the appearance of 1 or more new lesions. Stable disease (SD): neither sufficient shrinkage for PR nor sufficient increase for PD taking as reference smallest sum of LD since treatment started.
Time Frame: Part 1 Baseline, every 6 weeks up to 6 months
Population: Per protocol (PP) population included participants who received at least 14 doses of bosutinib and at least 10 doses of capecitabine within a 21-day period, had a baseline and at least 1 post-baseline tumor assessment, and had no major protocol violations.
Measure: Number; unit: Participants
Arm/Group | Bosutinib 200 mg + Capecitabine 625 mg/m^2 (Part 1) | Bosutinib 200 mg + Capecitabine 750 mg/m^2 (Part 1) | Bosutinib 200 mg + Capecitabine 1000 mg/m^2 (Part 1) | Bosutinib 300 mg + Capecitabine 625 mg/m^2 (Part 1) | Bosutinib 300 mg + Capecitabine 750 mg/m^2 (Part 1) | Bosutinib 300 mg + Capecitabine 1000 mg/m^2 (Part 1) | Bosutinib 400 mg + Capecitabine 750 mg/m^2 (Part 1) | Bosutinib 400 mg + Capecitabine 1000 mg/m^2 (Part 1)
Number analyzed (Participants) | 1 | 4 | 4 | 5 | 4 | 9 | 2 | 1
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Stable Disease | 0 | 1 | 2 | 0 | 1 | 6 | 1 | 1
  Progressive Disease | 1 | 3 | 2 | 5 | 1 | 2 | 1 | 0
  Indeterminate | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

5. Secondary Outcome: Progression Free Survival (PFS) - Part 2
Description: Time in weeks from randomization to first documentation of objective tumor progression or death due to any cause. PFS was calculated as (first event date minus the date of randomization plus 1) divided by 7. Tumor progression was determined from oncologic assessment data (where data meet the criteria for PD), or from adverse event (AE) data (where the outcome was "Death").
Time Frame: Part 2 Baseline, every 6 weeks up to 2 to 6 weeks after last dose
Population: as for outcome 3
Arm/Group | Bosutinib 300 mg + Capecitabine 1000 mg/m^2 (Part 2): ER+ | Bosutinib 300 mg + Capecitabine 1000 mg/m^2 (Part 2): ER-
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Clinical Benefit Rate - Part 2
Description: Percent of participants with confirmed CR, PR or SD for at least 24 weeks on study according to RECIST. CR: disappearance of all lesions. PR: at least 30% decrease in sum of LDs of target lesions taking as reference baseline sum LDs. SD: neither sufficient shrinkage for PR nor sufficient increase for PD taking as reference smallest sum of LD since treatment started.
Time Frame: Part 2 Baseline, every 6 weeks up to 2 to 6 weeks after last dose
Population: as for outcome 3
Arm/Group | Bosutinib 300 mg + Capecitabine 1000 mg/m^2 (Part 2): ER+ | Bosutinib 300 mg + Capecitabine 1000 mg/m^2 (Part 2): ER-
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Duration of Response (DR) - Part 2
Description: Time in weeks from the first documentation of objective tumor response to objective tumor progression or death due to any cancer. Duration of tumor response was calculated as (the date of the first documentation of objective tumor progression or death due to cancer minus the date of the first CR or PR that was subsequently confirmed plus 1) divided by 7. DR was calculated for the subgroup of participants with a confirmed objective tumor response.
Time Frame: Part 2 Baseline, every 6 weeks up to 2 to 6 weeks after last dose
Population: as for outcome 3
Arm/Group | Bosutinib 300 mg + Capecitabine 1000 mg/m^2 (Part 2): ER+ | Bosutinib 300 mg + Capecitabine 1000 mg/m^2 (Part 2): ER-
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) - Part 2
Time Frame: 0 hour (Pre-dose) on Day 1 and 2, 3, 4, 6, 8 and 24 hours post-dose on Day 14 of Cycle 1
Population: as for outcome 3
Arm/Group | Bosutinib 300 mg + Capecitabine 1000 mg/m^2 (Part 2): ER+ | Bosutinib 300 mg + Capecitabine 1000 mg/m^2 (Part 2): ER-
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) - Part 2
Time Frame: 0 hour (Pre-dose) on Day 1 and 2, 3, 4, 6, 8 and 24 hours post-dose on Day 14 of Cycle 1
Population: as for outcome 3
Arm/Group | Bosutinib 300 mg + Capecitabine 1000 mg/m^2 (Part 2): ER+ | Bosutinib 300 mg + Capecitabine 1000 mg/m^2 (Part 2): ER-
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Apparent Volume of Distribution (Vz/F) - Part 2
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: 0 hour (Pre-dose) on Day 1 and 2, 3, 4, 6, 8 and 24 hours post-dose on Day 14 of Cycle 1
Population: as for outcome 3
Arm/Group | Bosutinib 300 mg + Capecitabine 1000 mg/m^2 (Part 2): ER+ | Bosutinib 300 mg + Capecitabine 1000 mg/m^2 (Part 2): ER-
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-24)] - Part 2
Description: AUC (0-24) = Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-24).
Time Frame: 0 hour (Pre-dose) on Day 1 and 2, 3, 4, 6, 8 and 24 hours post-dose on Day 14 of Cycle 1
Population: as for outcome 3
Arm/Group | Bosutinib 300 mg + Capecitabine 1000 mg/m^2 (Part 2): ER+ | Bosutinib 300 mg + Capecitabine 1000 mg/m^2 (Part 2): ER-
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Apparent Oral Clearance (CL/F) - Part 2
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: 0 hour (Pre-dose) on Day 1 and 2, 3, 4, 6, 8 and 24 hours post-dose on Day 14 of Cycle 1
Population: as for outcome 3
Arm/Group | Bosutinib 300 mg + Capecitabine 1000 mg/m^2 (Part 2): ER+ | Bosutinib 300 mg + Capecitabine 1000 mg/m^2 (Part 2): ER-
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Terminal-Phase Disposition Rate Constant (λz) - Part 2
Description: The terminal-phase disposition rate constant measured by a log-linear regression of the terminal mono exponential portion of the observed plasma concentrations.
Time Frame: 0 hour (Pre-dose) on Day 1 and 2, 3, 4, 6, 8 and 24 hours post-dose on Day 14 of Cycle 1
Population: as for outcome 3
Arm/Group | Bosutinib 300 mg + Capecitabine 1000 mg/m^2 (Part 2): ER+ | Bosutinib 300 mg + Capecitabine 1000 mg/m^2 (Part 2): ER-
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Plasma Decay Half-Life (t1/2) - Part 2
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half. Half-life was to be calculated as 0.693/λz.
Time Frame: 0 hour (Pre-dose) on Day 1 and 2, 3, 4, 6, 8 and 24 hours post-dose on Day 14 of Cycle 1
Population: as for outcome 3
Arm/Group | Bosutinib 300 mg + Capecitabine 1000 mg/m^2 (Part 2): ER+ | Bosutinib 300 mg + Capecitabine 1000 mg/m^2 (Part 2): ER-
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Bosutinib 200 mg + Capecitabine 625 mg/m^2 (Part 1) | Bosutinib 200 mg + Capecitabine 750 mg/m^2 (Part 1) | Bosutinib 200 mg + Capecitabine 1000 mg/m^2 (Part 1) | Bosutinib 300 mg + Capecitabine 625 mg/m^2 (Part 1) | Bosutinib 300 mg + Capecitabine 750 mg/m^2 (Part 1) | Bosutinib 300 mg + Capecitabine 1000 mg/m^2 (Part 1) | Bosutinib 400 mg + Capecitabine 750 mg/m^2 (Part 1) | Bosutinib 400 mg + Capecitabine 1000 mg/m^2 (Part 1)
Serious Adverse Events (participants affected / at risk) | 0/2 | 2/4 | 2/4 | 2/5 | 0/4 | 3/9 | 0/2 | 1/2
Other Adverse Events (participants affected / at risk) | 2/2 | 4/4 | 3/4 | 5/5 | 4/4 | 9/9 | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bosutinib 200 mg + Capecitabine 625 mg/m^2 (Part 1) (N=2) | Bosutinib 200 mg + Capecitabine 750 mg/m^2 (Part 1) (N=4) | Bosutinib 200 mg + Capecitabine 1000 mg/m^2 (Part 1) (N=4) | Bosutinib 300 mg + Capecitabine 625 mg/m^2 (Part 1) (N=5) | Bosutinib 300 mg + Capecitabine 750 mg/m^2 (Part 1) (N=4) | Bosutinib 300 mg + Capecitabine 1000 mg/m^2 (Part 1) (N=9) | Bosutinib 400 mg + Capecitabine 750 mg/m^2 (Part 1) (N=2) | Bosutinib 400 mg + Capecitabine 1000 mg/m^2 (Part 1) (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bosutinib 200 mg + Capecitabine 625 mg/m^2 (Part 1) (N=2) | Bosutinib 200 mg + Capecitabine 750 mg/m^2 (Part 1) (N=4) | Bosutinib 200 mg + Capecitabine 1000 mg/m^2 (Part 1) (N=4) | Bosutinib 300 mg + Capecitabine 625 mg/m^2 (Part 1) (N=5) | Bosutinib 300 mg + Capecitabine 750 mg/m^2 (Part 1) (N=4) | Bosutinib 300 mg + Capecitabine 1000 mg/m^2 (Part 1) (N=9) | Bosutinib 400 mg + Capecitabine 750 mg/m^2 (Part 1) (N=2) | Bosutinib 400 mg + Capecitabine 1000 mg/m^2 (Part 1) (N=2)
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 2 | 3 | 3 | 8 | 2 | 2
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 4 | 2 | 2 | 1 | 4 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 3 | 1 | 0 | 1 | 2 | 2 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 1 | 3 | 1 | 5 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1 | 0 | 3 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 2 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 1 | 1 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0 | 1 | 3 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1

LIMITATIONS AND CAVEATS:
Results are not provided because the study was terminated prior to part 2 due to unfavorable risk benefit ratio of the study treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.